CLINICAL TRIAL: NCT05522218
Title: Clinical Effectiveness and Health Economic Evaluation of Eluvia Drug-eluting Stent in the Treatment of Femoropopliteal Artery Lesions
Brief Title: Eluvia DES for the Patients with Femoropopliteal Artery Lesions.
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Ziheng Wu, MD, Associated chief physician, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20220166B-X1
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Vascular Diseases; Stent Complication
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Eluvia drug eluting stent — Eluvia drug eluting stent for peripheral arterial disease

SUMMARY:
This study is a multicenter, prospective, observational study, aiming to enroll 400 patients with peripheral arterial disease in the femoral-popliteal segment implanted with Eluvia stent. Each patient was followed up for 2 years. The technical success rate, target lesion patency rate, quality of life improvement, cost of Eluvia stent implantation, and other outcomes will be analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Rutherford Stage 2-5.
2. At least 90% stenosis or occlusion of the femoropopliteal artery.
3. Eluvia stents are used for target lesions.
4. Agree and sign the informed consent form

Exclusion Criteria:

1. Life expectancy is less than 1 year.
2. Those with severe infection and gangrene of the limbs or those with tissue defects beyond the plane of the toes (ie major tissue loss), who may undergo major amputation even if the blood vessels are opened.
3. Patients and their families are reluctant to join the observational study, or have difficulty in communication and are unable to assess the quality of life.
4. Patients with in-stent restenosis of the femoral popliteal artery.
5. Patients with acute arterial thrombosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: peripheral arterial disease patients implanted with Eluvia stent
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of Rutherfor classification | 24 months
  Comparison of preoperative Rutherford classification and postoperative Rutherford classification at 24 months
F-TLR | 24 months
  free of target vascular reconstruction
limb salvage rate | 24 months
  Proportion of patients without ambutation

SECONDARY OUTCOMES:
Technical success rate | 1 month
  Percentage of patients with successful endovascular treatment without postoperative complications
the patency target lesion | 24 months
  Restenosis was defined as PSVR > 2.4 as determined by vascular ultrasonography
mortality rate | 24 months
  the propotion of death
the life quality change | 24 months
  Amount by Vas-Qol questionare between perioperation and 24month postoperation
the life quality change | 24 months
  Amount by EQ-5D5L questionare between perioperation and 24month postoperation
Economics Evaluation | 24 months
  Cumulative hospitalization expenses related to treatment within 24 months
Wound Healing Evaluation | 24 months
  If there is an ulcer wound, evaluate the ulcer wound healing at 24 months after surgery and before treatment

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
After recruitment, data will be shared after 2 years of follow-up